CLINICAL TRIAL: NCT04420572
Title: Comparison of Ozone and Steroid Injection in Patients With Greater Trochanteric Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Adem Erbirol
Record Dates: First submitted 2020-06-02; First posted 2020-06-09 (Actual); Results first posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Trochanteric Bursitis
Keywords: trochanteric bursitis; ozone; steroid; injection
MeSH Terms: interventions — Ozone; Betamethasone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ozone injection group (Experimental): ozone injection will be applied in three doses (1st, 4th, 7th and 10th days) for a total of 4 doses. In ozone injection applications, 1st dose 25 gamma, 2nd dose 20 gamma, 3rd and 4th dose 15 gamma 10 cc ozone will be injected.
  Interventions: Drug: ozone injection
- steroid injection group (Experimental): 1ml betamethasone will be used for steroid injection.
  Interventions: Drug: betamethasone

INTERVENTIONS:
Drug: ozone injection — ozone injection will be applied in three doses (1st, 4th, 7th and 10th days) for a total of 4 doses. In ozone injection applications, 1st dose 25 gamma, 2nd dose 20 gamma, 3rd and 4th dose 15 gamma 10 cc ozone will be injected.
  Other Names: no other names
  Arms: ozone injection group
Drug: betamethasone — 1ml betamethasone will be used for steroid injection.
  Other Names: no other names
  Arms: steroid injection group

SUMMARY:
Between the large trochanter and the muscles adhering to it, trochanteric bursa and several other bursa may be found. Trochanteric bursitis can be alone or together with tendinitis of other bursa and adhering muscles. The first is called trochanteric bursitis, the second is called hip periarthritis, which is difficult to distinguish clinically. It is more common in women of middle age. The main complaint is the large trochanter and pain on the side of the thigh. Pain is aggregated by walking abduction and external rotation by walking, lying down with hip movements. The palpation is sensitive to the top of the large trochanter. There may also be tenderness in the muscles in the lateral of the thigh. On plain radiographs, slight irregularities or peritrocanteric calcifications can be seen in the large trochanter. Bone scintigraphy shows local increased involvement. In differential diagnosis, stress fractures, local infection and bone and soft tissue tumors should be considered.

Rest is recommended in treatment. Activities such as running, standing for a long time are prohibited. Ice application can be given in the acute period. Non-steroidal anti-inflammatory (SOAI) drugs, analgesics, TENS can be used for pain relief. In cases where conventional treatments are insufficient, that is, the patient's pain is still continuing and functional recovery is inadequate, some alternative methods are also applied. These treatments include ozone, prolotherapy injection applications, dry needling, acupuncture, hirudotherapy, phytotherapy, mesotherapy, balneotherapy, kinesiobanding, etc. d. In our study, we aim to compare the effectiveness of ozone injection in patients diagnosed with trochanteric bursitis and to compare steroid injection with the application of ozone therapy.

DETAILED DESCRIPTION:
60 patients with trochanteric bursitis will be taken to the first and second groups by random number generator method. Ozone therapy is planned for 30 patients in the first group, and steroid injection is planned for the second group in 30 patients, and the study period is planned to be 4.5 months. Patients between the ages of 18-75 will be admitted and no difference will be made in terms of gender. The child will not be sick. Patients will be evaluated by the doctor who made the injection. All patients will also be evaluated before the first injection (T0), after treatment (T1) and after the first month (T2) after treatment. VAS (visual analog scale), Nottingham Health Profile and Harris Hip Evaluation Form will be used to evaluate patients. Our study is a randomized controlled prospective study.

Treatment to be applied to patients will be selected randomly. Steroid injections will be administered to patients in a single dose, while ozone injection will be applied in three doses (1, 4, 7, 10 days), with a total of 4 doses. In ozone injection applications, while 1st dose 25 gamma, 2nd dose 20 gamma, 3rd and 4th dose 15 gamma 10 cc ozone will be injected; 1ml betamethasone will be used for steroid injection. The evaluation of the patients will be done by a different physician than the physician who made the injections. The financial burden of the treatment applied will be borne by the researchers.

This study is a randomized controlled prospective clinical trial. The sample size is 60 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years of age, under 75 years of age
2. Lateral hip pain
3. Having pain for at least 3 months
4. The VAS value should be minimum 4 and pain is increased by pressing on t.major.
5. Conservative treatment failure

Exclusion Criteria:

1. Motor and / or sensory impairment compatible with radiculopathy
2. Connective tissue disease
3. Pregnancy
4. Active infection, immune system disorders, unresolved fractures
5. Hip op history, bursectomy / ilio-tibial band elongation
6. Steroid injection history in the past 4 months
7. Physical therapy history for trochanteric bursitis in the last 4 months
8. Rheumatological patients, pregnancy, Patients with a history of cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ADEM ERBİROL, Study Director — sultan abdulhamid han
Locations (1):
- Sultan 2.Abdülhamid Han Training and Research Hospital, Istanbul, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
other researchers would get information from the main researcher. therefore it was not shared.

RESULTS

PARTICIPANT FLOW:
Groups:
- Ozone Injection Group: The patients in the OI group received injections on the 1st, 4th, 7th and 10th days. A gas mixture containing 10 cc of 5% O3 and 95% medical O2 at a concentration of 25 μg/ml in the first application, 20 μg/ml in the second application, and 15 μg/ml in the third and fourth applications was used. It was the same physician who prepared and administered ozone. Experience has shown that a single dose of ozone application is not sufficient, it must be applied in sessions for a strong effect. Therefore, we used 4 doses of OI instead of a single dose in our study
- Steroid Injection Group: A single dose injection was given to the patients in the CSI group. The solution to be administered to the CSI group was obtained by mixing 1 ml of 2% lidocaine and 1 ml of betamethasone (Diprospan 2 mg/1ml+5 mg/1ml). It was the same physician who prepared and administered the solutions. In the studies, it was generally applied as a single dose and mixed with local anesthetic (LA). Therefore, in our study, we also applied it as a single dose by mixing it with LA.
Period: Overall Study
Arm/Group | Ozone Injection Group | Steroid Injection Group
Started | 33 | 30
Completed | 33 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ozone Injection Group: The patients in the ozone injection (OI) group received injections on the 1st, 4th, 7th and 10th days. A gas mixture containing 10 cc of 5% O3 and 95% medical O2 at a concentration of 25 μg/ml in the first application, 20 μg/ml in the second application, and 15 μg/ml in the third and fourth applications was used. It was the same physician who prepared and administered ozone. Experience has shown that a single dose of ozone application is not sufficient, it must be applied in sessions for a strong effect. Therefore, we used 4 doses of OI instead of a single dose in our study.
- Steroid Injection Group: A single dose injection was given to the patients in the corticosteroids (CSI) group. The solution to be administered to the CSI group was obtained by mixing 1 ml of 2% lidocaine and 1 ml of betamethasone (Diprospan 2 mg/1ml+5 mg/1ml). It was the same physician who prepared and administered the solutions. In the studies, it was generally applied as a single dose and mixed with local anesthetic (LA). Therefore, in our study, we also applied it as a single dose by mixing it with LA.
- Total: Total of all reporting groups
Arm/Group | Ozone Injection Group | Steroid Injection Group | Total
Number analyzed (Participants) | 33 | 30 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 23 | 49
  >=65 years | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.85 (11.82) | 54.87 (12.95) | 54.33 (12.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 26 | 54
  Male | 5 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 33 | 30 | 63
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 33 | 30 | 63
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.68 (4.41) | 29.64 (4.37) | 29.14 (4.38)

OUTCOME MEASURES:

1. Primary Outcome: Pain Severity
Description: visual analog scale (0-10) minimum score: 0 maximum score: 10. Higher scores reflect more severe pain
Time Frame: day 0 (before intervention)
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ozone Injection Group | Steroid Injection Group
Number analyzed (Participants) | 33 | 30
score on a scale | 8.36 (1.06) | 8.17 (0.95)

2. Primary Outcome: Pain Severity
Description: visual analog scale (0-10) minimum score: 0 maximum score: 10. Higher scores reflect more severe pain
Time Frame: 1 week after intervention
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ozone Injection Group | Steroid Injection Group
Number analyzed (Participants) | 33 | 30
score on a scale | 3.64 (2.28) | 2.93 (2.27)

3. Primary Outcome: Pain Severity
Description: visual analog scale (0-10) minimum score: 0 maximum score: 10. Higher scores reflect more severe pain
Time Frame: 1 month after intervention
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ozone Injection Group | Steroid Injection Group
Number analyzed (Participants) | 33 | 30
score on a scale | 3.30 (3.15) | 3.00 (2.41)

4. Secondary Outcome: Functionality
Description: harris hip score: gives information about the functionality of patients. harris hip score minimum score: 0 maximum score: 100. High scores reflect better functionality
Time Frame: day 0 (before intervention)
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ozone Injection Group | Steroid Injection Group
Number analyzed (Participants) | 33 | 30
score on a scale | 53.03 (5.87) | 53.03 (5.97)

5. Secondary Outcome: Functionality
Description: as for outcome 4
Time Frame: 1 week after intervention
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ozone Injection Group | Steroid Injection Group
Number analyzed (Participants) | 33 | 30
score on a scale | 72.85 (12.02) | 75.00 (7.56)

6. Secondary Outcome: Functionality
Description: as for outcome 4
Time Frame: 1 month after intervention
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ozone Injection Group | Steroid Injection Group
Number analyzed (Participants) | 33 | 30
score on a scale | 72.79 (12.58) | 74.97 (6.89)

7. Secondary Outcome: Patient Reported Quality of Life - Notthingham Health Profile
Description: Notthingham Health Profile: general patient reported outcome measure which measures subjective health status.
  38 questions in 6 subareas, with each question assigned a weighted value; the sum of all weighted valuesin a given subarea adds up to 100. Overall score is calculated by summing up 6 subdomian scores.
  Overall minimum: 0 maximum: 600 (6X100) Higher scores reflect worse health status
Time Frame: day 0 (before intervention)
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ozone Injection Group | Steroid Injection Group
Number analyzed (Participants) | 33 | 30
score on a scale | 261.72 (109.77) | 255.51 (127.22)

8. Secondary Outcome: Patient Reported Quality of Life - Notthingham Health Profile
Description: as for outcome 7
Time Frame: 1 week after intervention
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ozone Injection Group | Steroid Injection Group
Number analyzed (Participants) | 33 | 30
score on a scale | 215.40 (106.58) | 193.04 (103.10)

9. Secondary Outcome: Patient Reported Quality of Life - Notthingham Health Profile
Description: as for outcome 7
Time Frame: 1 month after intervention
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ozone Injection Group | Steroid Injection Group
Number analyzed (Participants) | 33 | 30
score on a scale | 210.28 (108.58) | 188.62 (109.10)

ADVERSE EVENTS:
Time Frame: adverse events were not monitored/assessed
Description: adverse events were not monitored/assessed
Arm/Group | Ozone Injection Group | Steroid Injection Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT04420572/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT04420572/SAP_001.pdf